CLINICAL TRIAL: NCT05154825
Title: Evaluating and Establishing the Relationship in the Five Critical X-ray Time Points in Spinal Deformity Realignment: Preoperative Standing and Supine, Intraoperative Pre- and Post-correction, and Postoperative Standing Films
Brief Title: Evaluating and Establishing the Relationship in the Five Critical X-ray Time Points in Spinal Deformity Realignment
Status: Recruiting | Type: Observational
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Joseph Osorio, Assistant Professor of Neurological Surgery, University of California, San Diego
Other Study IDs: 210830
Record Dates: First submitted 2021-11-10; First posted 2021-12-13 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-05

CONDITIONS: Spine; Spine Deformity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Spine Surgery Participants: Spine surgical candidates that will be receiving posterior only surgery for spinal deformity
  Interventions: Other: Imaging-Observational

INTERVENTIONS:
Other: Imaging-Observational — Preoperative standing and supine, intraoperative pre- and post-correction, and postoperative standing imaging as well as imaging collected during follow-up exams for a year following surgery

SUMMARY:
To establish the relationship in the five critical X-ray time points during multilevel posterior column osteotomies (MPCO) spinal deformity realignment in patients with adult spinal deformity and to follow the participants longitudinally to examine any follow-up X-rays and clinical data to compare to the post-operative standing scan and pre-operative data.

DETAILED DESCRIPTION:
Studies in adult spinal deformity (ASD) have found that the presence of sagittal imbalance directly correlates with worsening quality of life. Multilevel posterior column osteotomies (MPCOs) is a technique that can provide correction to adult spinal deformity. MPCOs can be utilized for revision surgery as an alternative to 3-column osteotomies and have the ability to aggregate large amount of lordosis segmentally. The success of the MPCO technique largely depends on radiographs taken during these surgeries to aid the surgeon in establishing the best screw and rod placement and making intraoperative adjustments. Imaging plays a vital role in evaluating hardware positioning and assessing hardware integrity as well as evaluating potential complication. The investigator plans to evaluate and establish the relationship in the five critical X-ray time points (preoperative standing and supine, intraoperative pre- and post-correction, and postoperative standing films) during MPCO spinal deformity realignment and measure pre- to post-operative outcome longitudinally. The investigator will investigate lumbar lordosis and sagittal and coronal alignment at those 5 time points and examine the relationship between pre-op, intra-op, and post-op images to understand impact of the MPCO technique and examine expected outcome to final outcome. Additionally, if the O-Arm 2D long film scanner is utilized during the surgery, the investigator will analyze that film and compare it to the other X-rays taken.

ELIGIBILITY:
Inclusion Criteria:

* Surgical Candidate for posterior only surgery for adult spinal deformity
* Patients must require deformity correction greater than 3 levels
* Adults Between the ages of 18-80
* Decisional capacity to consent to the study
* Both Primary and revision surgeries will be included

Exclusion Criteria:

* 1) Not meeting candidacy for posterior spine surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The cohort will be select from the UCSD Neurological Surgery Spine clinic who are candidates for Posterior Spinal Surgery involving more then 3 levels of posterior column osteotomies
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2021-12-07 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Evaluate the Change from Baseline Sagittal Cobb angles to Post-Surgical Sagittal Cobb angles | Baseline through end of Hospital Stay, an average of 6 weeks
  Data analysis will involve analysis of the change of segmentally measured Sagittal Cobbs angles in the presurgical baseline, intra-operative and post-surgical X-rays
Evaluate the Change from Baseline Total Lumbar Lordosis to Post-Surgical Total Lumbar Lordosis | Baseline through end of Hospital Stay, an average of 6 weeks
  Data analysis will involve analysis of the change of measured total lumbar lordosis in the presurgical baseline, intra-operative and post-surgical X-rays

SECONDARY OUTCOMES:
Evaluation of the change of Sagittal Cobb angles in post-operative X-rays taken at follow-up appointments for the first year post surgery | Through study completion, an average of 1 year
  Data analysis will involve analysis of the post-surgical X-rays utilizing the Sagittal Cobb angles measured segmentally
Evaluation of the change of total lumbar lordosis in post-operative X-rays taken at follow-up appointments for the first year post surgery | Through study completion, an average of 1 year
  Data analysis will involve analysis of the post-surgical X-rays utilizing the angle for lumbar lordosis

OTHER OUTCOMES:
PROMIS-29 (Patient-Reported Outcomes Measurement Information System-29 question) questionnaire | Through study completion, an average of 1 year
  The PROMIS-29 will be given to assess change over time in global physical, mental and social health.
Oswestry Disability Index | Through Study Completion, an average of 1 year
  The Oswestry Disability Index will be given to assess change over time in functional disability
SRS-22r (Scoliosis Research Society Patient Outcome Questionnaire) | Through Study Completion, an average of 1 year
  The SRS-22r (Scoliosis Research Society Patient Outcome Questionnaire) will be given to assess change in the health related quality of life specific to spinal deformity
Visual Analog Scale (VAS) Low Back and/or Leg | Through Study Completion, an average of 1 year
  The Visual Analog Scale (VAS) for Low Back and/or Leg will be given to assess changes in pain level.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Osorio, MD, PhD, Principal Investigator — University of California, San Diego
Locations (1):
- University of California, San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Undecided
Sharing of IPD depends on future relevant collaborations that require IPD to be shared

REFERENCES:
- [Background] Chan AK, Lau D, Osorio JA, Yue JK, Berven SH, Burch S, Hu SS, Mummaneni PV, Deviren V, Ames CP. Asymmetric Pedicle Subtraction Osteotomy for Adult Spinal Deformity with Coronal Imbalance: Complications, Radiographic and Surgical Outcomes. Oper Neurosurg. 2020 Feb 1;18(2):209-216. doi: 10.1093/ons/opz106. PMID 31214712
- [Background] Scheer JK, Osorio JA, Smith JS, Schwab F, Hart RA, Hostin R, Lafage V, Jain A, Burton DC, Bess S, Ailon T, Protopsaltis TS, Klineberg EO, Shaffrey CI, Ames CP; International Spine Study Group. Development of a Preoperative Predictive Model for Reaching the Oswestry Disability Index Minimal Clinically Important Difference for Adult Spinal Deformity Patients. Spine Deform. 2018 Sep-Oct;6(5):593-599. doi: 10.1016/j.jspd.2018.02.010. PMID 30122396
- [Background] Lau D, Osorio JA, Deviren V, Ames CP. The relationship of older age and perioperative outcomes following thoracolumbar three-column osteotomy for adult spinal deformity: an analysis of 300 consecutive cases. J Neurosurg Spine. 2018 Jun;28(6):593-606. doi: 10.3171/2017.10.SPINE17374. Epub 2018 Apr 6. PMID 29624129